CLINICAL TRIAL: NCT00177229
Title: Family-Based Treatment of Severe Pediatric Obesity
Brief Title: KidQuest Family-Based Weight Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Marsha D. Marcus, Ph.D., Professor of Psychiatry, University of Pittsburgh School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0405048
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (No Intervention): Enhanced usual care: 2 free, individual consultations with a nutritionist over first 6 months. Medical monitoring throughout study period.
- B (Experimental)
  Interventions: Behavioral: Family-based treatment

INTERVENTIONS:
Behavioral: Family-based treatment — 20 weekly group contacts with individual coaching over first 6 months, brief monthly contacts over next 6 months, no contacts over last 6 months. Medical monitoring throughout study period.
  Arms: B

SUMMARY:
The purpose of this study is to determine if a family based diet and exercise program is helpful for extremely overweight children aged 8-12, and to compare this approach to standard medical management of severe pediatric obesity.

DETAILED DESCRIPTION:
The prevalence of pediatric obesity has increased significantly, and approximately 11% of American children and adolescents are obese. Of particular concern, the greatest increase in prevalence has occured among the heaviest children. Severe pediatric obesity (defined as > 150% of ideal body weight for height) is associated with higher rates of medical and psychosocial morbidity than milder obesity is. Moreover, severely obese children are likelier than less severely obese children are to become obese adults and suffer the long-term health consequences of obesity. Although the efficacy of family-based behavioral weight control programs in the treatment of moderate pediatric obesity is well established, few studies have focused on the treatment of severe obesity. Thus in this application, we propose a randomized controlled trial to evaluate the efficacy of a family-based behavioral weight control program in the management of severe pediatric obesity.

Two hundred children aged 8-12 will be randomized to a six-month family-based program or usual care, and will complete assessments at pre- and post- treatment and 6-month and 12-month follow-ups. We hypothesized that: 1) Children who participate in the family-based program, when compared to children who receive usual care, will show favorable changes in body mass index, body composition, food intake, activity level, and cardiovascular risk factors. 2) Children who participate in the family-based program, when compared to children who receive usual care, will report higher levels of self-esteem, social competence and health-related quality of life, and report fewer psychiatric symptoms. A secondary aim of the the proposed investigation is to examine the relationships among gender, race, compliance to diet and exercise. level of parent adherence and treatment outcome. The proposed investigation is significant as the first effort to systematically evaluate a treatment program for severely obese children. It will provide data about a serious public health problem and establish a foundation for programmatic research to develop effective treatments for an underserved population.

ELIGIBILITY:
Inclusion Criteria:

* Be >150% of ideal body weight for height and age based on norms of the World Health Organization.
* Have at least one parent or guardian who will participate in the treatment program with child.

Exclusion Criteria:

* Mental retardation, pervasive developmental disorder or psychosis, psychiatric symptomatology sufficiently severe to require immediate treatment.
* Genetic obesity syndrome as determined by the study physician.
* Currently receiving obesity treatment and/or participating in a weight management program.
* Inability to engage in moderate exercise defined as 30 minutes of vigorous activity on most days of the week.
* Acute or severe medical conditions that require aggressive weight management intervention (e.g., diabetes pseudotumor cerebri, or hypoventilation).
* Regular use of a medication that affects body weight such as oral steroids or antipsychotic medications.
* Taking stimulant or antidepressant medication for a period < four months.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2001-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
BMI and cardiovascular risk factors | 0,6,12,18

SECONDARY OUTCOMES:
Eating, activity, and psychosocial functioning | 0,6,12,18

CONTACTS AND LOCATIONS:
Overall Officials: Marsha D. Marcus, Ph.D., Principal Investigator — Western Psychiatric Insitute & Clinic